CLINICAL TRIAL: NCT01186718
Title: Three-dimensional Study of Cervical Kinematics
Brief Title: Interexaminer Reliability, Outcomes for Manipulation of Cervical Dysfunction, 3-D Kinematics
Status: Completed | Type: Observational
Sponsor: Michigan State University (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Principal Investigator, Joseph Vorro, Professor and PI, Michigan State University
Other Study IDs: AOA 09-05-581
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Human Cervical Motions
Keywords: Cervical, motions, kinematics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control Group: Control group = functional symmetric cervical motion.
- Experimental subject group: Experimental subject group = asymmetric cervical motion

SUMMARY:
The purpose of this project is to quantify 3-dimensional (3-D) cervical motion pattern changes that result from osteopathic manipulation treatment (OMT) in an experimental subject group diagnosed with somatic dysfunction. The kinematic data will include the entire 3-D motion trajectories of the head, resulting in range of motion (ROM) and angular data for the primary and secondary motions.

DETAILED DESCRIPTION:
Our primary hypothesis is that kinematic changes will be detected after OMT for motions in the primary direction of the passive diagnostic test motions (cervical side-bending right and left), as well as angular rotations (deviations) occurring around these motions. Our secondary hypothesis is that examination of the kinematic data will provide objective inter- and intra-examiner data to assess similarities/differences occurring during the passive clinical exam before and after OMT. Lastly, we hypothesize that significant differences in the kinematic patterns will result between the two subject groups.

This experiment is designed for the following clinical and biomechanical observations:

* comparisons of diagnostic data between three osteopathic physicians,
* comparisons of within-subject kinematic profiles pre- and post-treatment,
* inter-examiner comparisons of kinematic motion paths occurring during diagnostic motions,
* evaluate kinematic patterns between the two subject groups, and assess between group similarities/differences,
* evaluate diagnostic and kinematic data relative to VAS, cervical disability, health status information, and SNF,
* re-classify aspects of the kinematic data using a cluster (statistical) analysis procedure to compare with initial and secondary physician diagnostic data, and
* to assess the stability of changes made by the OMT procedures and the kinematic response three days post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Cervical motion symmetry and asymmetry

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two study groups: Control = subjects with symmetric cervical motion; Experimental = subjects with asymmetric cervical motion.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
3-D kinematic measurements of cervical motion | 9/2009 to 8/2011

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Vorro, Phd, Principal Investigator — Michigan State University Dept. Family Medicine
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

REFERENCES:
- [Derived] Vorro J, Bush TR, Rutledge B, Li M. Kinematic measures during a clinical diagnostic technique for human neck disorder: inter- and intraexaminer comparisons. Biomed Res Int. 2013;2013:950719. doi: 10.1155/2013/950719. Epub 2013 Feb 16. PMID 23509819